CLINICAL TRIAL: NCT02219581
Title: Evaluation of Intravenous Glucocorticoid Therapy in Total Knee Arthroplasty
Brief Title: Steroids in Total Knee Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated after considerable time in suspended state due to inadequate staffing, the COVID pandemic, and the Responsible Party leaving Emory in August 2022.
Sponsor: Thomas L Bradbury (Other)
Responsible Party: Sponsor-Investigator, Thomas L Bradbury, Associate Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00066081
Record Dates: First submitted 2014-08-13; First posted 2014-08-19 (Estimated); Results first posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Pain; Inflammation; Osteoarthritis
Keywords: Osteoarthritis; Postoperative pain; Total knee arthroplasty; Orthopaedics; Inflammation
MeSH Terms: conditions — Pain, Postoperative; Inflammation; Osteoarthritis | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects undergoing primary total joint arthroplasty of the knee will receive two doses of placebo intravenously in addition to a standard multimodal postoperative pain management regimen typically used for total knee arthroplasty. The first dose of placebo will be given preoperatively within 3 hours of surgery and the second dose will be administered 8 hours after the first dose in the inpatient setting.
  Interventions: Drug: Standard multimodal pain management regimen; Drug: Placebo
- Dexamethasone 10 mg (Experimental): Subjects undergoing primary total joint arthroplasty of the knee will receive two doses of 10 mg dexamethasone. The first dose will be given preoperatively within 3 hours of surgery and the second dose will be administered 8 hours after the first dose in the inpatient setting. Additionally, subjects will also receive a standard multimodal postoperative pain management regimen typically used for total knee arthroplasty.
  Interventions: Drug: Dexamethasone 10 mg; Drug: Standard multimodal pain management regimen
- Dexamethasone 20 mg (Experimental): Subjects undergoing primary total joint arthroplasty of the knee will receive two doses of 20 mg dexamethasone. The first dose will be given preoperatively within 3 hours of surgery and the second dose will be administered 8 hours after the first dose in the inpatient setting. Additionally, subjects will also receive a standard multimodal postoperative pain management regimen typically used for total knee arthroplasty.
  Interventions: Drug: Dexamethasone 20 mg; Drug: Standard multimodal pain management regimen

INTERVENTIONS:
Drug: Dexamethasone 10 mg — Two doses of dexamethasone 10 mg will be given intravenously. The first dose will be given preoperatively within 3 hours of surgery and the second dose will be administered 8 hours after the first dose in the inpatient setting.
  Other Names: Decadron
  Arms: Dexamethasone 10 mg
Drug: Dexamethasone 20 mg — Two doses of dexamethasone 20 mg will be given intravenously. The first dose will be given preoperatively within 3 hours of surgery and the second dose will be administered 8 hours after the first dose in the inpatient setting.
  Other Names: Decadron
  Arms: Dexamethasone 20 mg
Drug: Standard multimodal pain management regimen — The standard multimodal postoperative pain management regimen typically used for total knee arthroplasty consists of the following:
  Preoperative:
  * Decadron: 10 or 20mg IV x 1 2 doses, 8 hours apart (if randomized to study group)
  Intraoperative:
  * Ropivacaine: Given intraoperatively. Capsule, subcutaneous tissue/skin. Administered in standard fashion. (300mg)
  * Toradol: 30mg q 6hr for 6 total doses. 1st dose given intraoperatively at incision. The dose is 15 mg for older patients or if creatinine clearance (CrCl) is low.
  Postoperative
  * Tylenol: 1000mg po q 8hr (scheduled)
  * Oxycodone: 5mg or 10mg q 3-4hr prn pain, If intolerant to Oxycodone: second agent line is Hydrocodone or Oral Dilaudid
  * IV Morphine (or Dilaudid): 1 or 2 mg q 2hr prn breakthrough pain
  * Morphine patient-controlled analgesia (PCA): only for failure of the above
  * Morphine Sulfate (MS) Contin: Use as backup prn pain
Drug: Placebo — Participants in the placebo arm will receive two doses of saline intravenously. The first dose will be given preoperatively within 3 hours of surgery and the second dose will be administered 8 hours after the first dose in the inpatient setting.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if the use of two small doses of intravenous (IV) steroids around the time of knee replacement surgery decrease a patient's pain or use of pain medication. The investigators will also determine if the subjects receiving the steroid will have better pain control and better postoperative outcomes after their surgery.

DETAILED DESCRIPTION:
Adequate pain control after total knee arthroplasty (TKA) is of great importance not only to maximize patient comfort, but also to ensure optimal outcomes after surgery. This study is designed to assess whether the use of two small doses of intravenous (IV) steroids around the time of surgery decrease a patient's pain or use of pain medication. Secondly, the investigators will also determine if the use of these steroids as part of a multimodal pain management strategy leads to improved patient outcomes, including pain, nausea and vomiting, knee function and length of stay in the hospital after surgery. The study will compare the effect of two different doses of IV dexamethasone given preoperatively before TKA, when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary total joint arthroplasty of the knee
* Adult patients ages 18-100 years
* Patients must have smart phone and/or device for app usage

Exclusion Criteria:

* Current chronic steroid use
* Patients undergoing revision knee surgery
* Patients ambulating preoperatively with assistive devices
* Patients with avascular necrosis of the operative knee
* Patients with a history of an adverse reaction to glucocorticoid steroids
* Patients unable to provide informed consent
* Patients with inflammatory arthritis
* Prisoners
* Current smokers
* Patients <18 years of age
* Any patient with a complicated postoperative course that requires transfer to the Intensive Care Unit (ICU) or to another facility for further management will be removed from the study.
* Any contraindication that would prevent the patient from being treated with the standard multimodal postoperative pain management regimen History of infection of surgical knee.
* Patients with diabetes.
* Patients that have an intolerance to Toradol.
* Patients that do not have smart phone and/or device for app usage

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Bradbury, MD, Principal Investigator — Emory University
Locations (1):
- Emory Orthopedic and Spine Hospital, Tucker, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants undergoing primary total joint arthroplasty of the knee who are randomized to receive two doses of placebo intravenously in addition to a standard multimodal postoperative pain management regimen typically used for total knee arthroplasty. The first dose of placebo will be given preoperatively within 3 hours of surgery and the second dose will be administered 8 hours after the first dose in the inpatient setting.
- Dexamethasone 10 mg: Participants undergoing primary total joint arthroplasty of the knee who are randomized to receive two doses of 10 mg dexamethasone. The first dose will be given preoperatively within 3 hours of surgery and the second dose will be administered 8 hours after the first dose in the inpatient setting. Additionally, participants will also receive a standard multimodal postoperative pain management regimen typically used for total knee arthroplasty.
- Dexamethasone 20 mg: Participants undergoing primary total joint arthroplasty of the knee who are randomized to receive two doses of 20 mg dexamethasone. The first dose will be given preoperatively within 3 hours of surgery and the second dose will be administered 8 hours after the first dose in the inpatient setting. Additionally, participants will also receive a standard multimodal postoperative pain management regimen typically used for total knee arthroplasty.
Period: Overall Study
Arm/Group | Placebo | Dexamethasone 10 mg | Dexamethasone 20 mg
Started | 0 | 0 | 1
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dexamethasone 20 mg: The participant undergoing primary total joint arthroplasty of the knee was randomized to receive two doses of 20 mg dexamethasone. The first dose was given preoperatively within 3 hours of surgery and the second dose was administered 8 hours after the first dose in the inpatient setting. Additionally, the participant received a standard multimodal postoperative pain management regimen typically used for total knee arthroplasty.
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: To maintain anonymity of the single participant of this study sex is not reported.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Post-operative pain was assessed using the well-standardized and accepted visual analog pain scale. The scale shows a series of faces ranging from a happy face at 0= "No hurt", to a crying face at 10= "Hurts worst". The participant was asked to choose the face that best describes their level of pain. Higher scores indicate higher intensities of pain.
Time Frame: Baseline, end of hospital stay (up to 3 days), 1, 4, and 12 months post-operatively
Measure: Number; unit: units on a scale
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 1
units on a scale
  Baseline | 3
  End of hospital stay (up to 3 days post-operative) | 0
  1 month post-operative | 0
  4 months post-operative | 3
  12 months post-operative | 0

2. Primary Outcome: Opioid Analgesic Usage
Description: The amount of post-operative opioid analgesic usage is assessed as Oral Morphine Equivalents (OME) which is the amount of an oral morphine drug that would be necessary to equal the pain treatment from opioid morphine.
Time Frame: 1 day post-operatively
Measure: Number; unit: Oral Morphine Equivalents (OME)
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 1
Oral Morphine Equivalents (OME) | 37.5

3. Secondary Outcome: Soft Tissue Swelling
Description: Evaluation of soft tissue swelling uses a measurement of knee circumference at the midpoint of the patella, with the knee in the maximum amount of extension allowed by the patient.
Time Frame: 1 day post-operatively
Population: Measurements of knee circumference were not obtained at any study time point, or measurements have been lost and are no longer available.
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 0

4. Secondary Outcome: Range of Motion (ROM)
Description: Maximum passive ROM allowed by the patient will be measured using a goniometer. The ROM measurement is the amount of flexion and extension recorded in degrees. An increased ROM is indicative of better joint mobility.
Time Frame: Baseline, 1 day post-operatively, 1, 4, and 12 months post-operatively
Measure: Number; unit: degrees
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 1
degrees
  Baseline | 125
  1 Day Post-Operative | 105
  1 Month Post-Operative | 135
  4 Months Post-Operative | 140
  12 Months Post-Operative | 110

5. Secondary Outcome: Post-operative Day of Physical Therapy Clearance
Description: The post-operative day when the participant was cleared by the physical therapy staff to go home was recorded. A shorter clearance time is indicative of better joint function.
Time Frame: Up to 3 days post-operatively
Measure: Number; unit: days
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 1
days | 3

6. Secondary Outcome: Antiemetic Dose Administered
Description: Post-operative nausea and/or vomiting was assessed by the use of the antiemetic Zofran, which was administered as-needed.
Time Frame: Post-operative Days 1 and 2
Measure: Number; unit: milligrams (mg)
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 1
milligrams (mg)
  Post-operative Day 1 | 4
  Post-operative Day 2 | 0

7. Secondary Outcome: Blood Glucose
Description: To assess postoperative glucose levels after steroid administration, blood glucose level will be analyzed using a HemoCue testing system. Diabetes is indicated with a random blood glucose measurement of greater than 200 milligrams per deciliter (mg/dL).
Time Frame: Baseline, Post-operative Day 1
Measure: Number; unit: mg/dL
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 1
mg/dL
  Baseline | 100
  Post-operative Day 1 | 88

8. Secondary Outcome: 36-Item Short Form Health Survey (SF-36) Score
Description: The subjects' functional ability will be assessed using the SF-36 questionnaire. The SF-36 Health Survey is a 36-item, self-reported survey of patient health and is a measure of health status. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The lower the score the more disability.
Time Frame: Baseline, 12 months post-operatively
Population: SF-36 scores are not available. The survey was either not administered or scores have been lost.
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 0

9. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) Score
Description: The KOOS, JR. instrument has 7 items assessing knee stiffness, knee pain, and daily living physical function following knee joint replacement. Responses are given on a 5-point scale where 0 = no pain or disability and 4 = extreme pain or disability. Total raw scores range from 0 to 28, where higher scores indicate increased pain or disability. Total raw scores can be converted to an interval score ranging from 0 to 100 where 0 = total knee disability and 100 = perfect knee health.
Time Frame: Baseline, 1, 4, and 12 months post-operatively
Population: KOOS, JR. scores are not available. The survey was either not administered or scores have been lost.
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 0

10. Secondary Outcome: Length of Hospital Stay
Description: The length of hospital stay in days is reported here. A higher number of days in the hospital indicates slower recovery.
Time Frame: Up to 3 days post-operatively
Measure: Number; unit: days
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 1
days | 3

11. Secondary Outcome: Number of Participants Readmitted to the Hospital
Description: The number of participants with hospital readmissions after being discharged were recorded.
Time Frame: Up to 12 months post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 1
Participants | 0

12. Secondary Outcome: Number of Participants With Wound Infections
Description: The number of participants with the clinical presence of wound drainage and periprosthetic infection were recorded.
Time Frame: Up to 12 months post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 20 mg
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from medical records beginning at the baseline assessment just prior to surgery and continued through the 12 month post-operative assessment (for 12 months total).
Arm/Group | Dexamethasone 20 mg
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
There are limitations of the study results due to termination of the study and a small number of study participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT02219581/Prot_SAP_000.pdf